CLINICAL TRIAL: NCT06307184
Title: Assessing the Convenience of Natural Proliferative Phase Frozen Embryo Transfer: an Ambispective Cohort Study
Brief Title: Assessing the Convenience of Natural Proliferative Phase Frozen Embryo Transfer
Status: Recruiting | Type: Observational
Sponsor: Instituto Valenciano de Infertilidade de Lisboa (Network)
Collaborators: Gedeon Richter Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2301-LIS-007-AN
Record Dates: First submitted 2024-02-17; First posted 2024-03-12 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Frozen Embryo Transfer
Keywords: Endometrial preparation; Natural cycle; Progesterone; Pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Natural proliferative phase frozen embryo transfer (NPP-FET): When the endometrial thickness is at least 7 mm, vaginal micronized progesterone will be initiated at 400mg every 12 hours, as per standard clinical practice, when the dominant follicle is at least 13 mm, serum estradiol (E2) levels are >80 pg/ml, and serum progesterone levels are <1.5ng/ml. One embryo will be transferred on the fifth day of progesterone supplementation under ultrasound guidance. Progesterone will be continued until the 11th week of pregnancy.
  Interventions: Procedure: Natural proliferative phase frozen embryo transfer
- Natural cycle frozen embryo transfer (NC-FET): When the mean dominant follicle diameter was at least 17 mm and the endometrial thickness was at least 7 mm, serum E2, progesterone and luteinizing hormone (LH) were evaluated. If a spontaneously LH peak was detected (E2>80 pg/ml, LH peak >18 mIU/mL with progesterone level <1.5 ng/mL), vaginal micronized progesterone was started from the evening of ovulation at a dose of 200 mg every 12 hours. Conversely, whenever a LH peak was not detected (E2>80 pg/ml, LH <18mIU/ml and progesterone <1,5 ng/ml), r-hCG 250µg (Ovitrelle®) was administered subcutaneously, followed, 48 hours later, by daily administration of 200 mg micronized vaginal progesterone every 12 hours. One embryo was transferred 7 days after r-hCG administration or 6 days after LH peak detection. Progesterone was continued until the 8th week of pregnancy.

INTERVENTIONS:
Procedure: Natural proliferative phase frozen embryo transfer — When endometrial thickness is above 7 mm, vaginal micronized progesterone will be administered 400mg 12/12h when the dominant follicle is at least 13 mm, serum estradiol (E2) levels are >80 pg/ml, and serum progesterone levels are <1.5ng/ml. Embryo transfer will be performed on the fifth day of progesterone.
  Groups: Natural proliferative phase frozen embryo transfer (NPP-FET)

SUMMARY:
This study will assess the convenience of the natural proliferative phase frozen embryo transfer (NPP-FET) in terms of number of number of appointments needed before cycle scheduling.

DETAILED DESCRIPTION:
Frozen embryo transfer (FET) is increasingly used nowadays in Assisted Reproductive Techniques (ART) clinics. Several factors account for this uprising. Among them, the concept of ovarian hyperstimulation syndrome (OHSS)-free clinic, the increasing use of preimplantation genetic testing (PGT), the improved vitrification systems, and the growing evidence regarding similar, or even better, pregnancy rates when FET are compared to fresh embryo transfers.

In the last few years, research has focused on the selection of the best protocol for endometrial preparation in patients undergoing FET cycles. Despite the accumulating evidence suggesting similar reproductive outcomes following both artificial cycle (AC-FET) and natural cycle (NC-FET) protocols, AC-FET is frequently adopted in ART centers due to its convenience in terms of cycle scheduling. However, a role for the corpus luteum in the maternal vasodilatory changes of early pregnancy has recently been associated with a decreased risk of pre-eclampsia. In fact, several large cohort studies have reported a higher risk of hypertensive diseases of pregnancy, macrosomia, post-term delivery and cesarean section following AC-FET.

The NPP-FET protocol is a strategy that potentially allows for cycle scheduling while maintaining the benefits of the natural cycle in terms of pregnancy outcomes. The main goal of the present study is to analyze its convenience in terms of the number of appointments needed before FET scheduling by comparing it with the NC-FET protocol. Additionally, the investigators aim to compare the reproductive outcomes between the two strategies and to analyze whether NPP-FET patients undergo ovulation.

Briefly, the study group will prospectively recruit ovulatory patients who will perform vaginal ultrasound monitoring will be performed on cycle day 8-12, depending on the length of the patients' menstrual cycle. When the endometrial thickness is at least 7 mm and the dominant follicle is at least 13 mm, vaginal micronized progesterone will be initiated at 400mg every 12 hours. One embryo will be transferred on the fifth day of progesterone supplementation under ultrasound guidance. The control group will include a retrospective cohort of ovulatory patients who underwent NC-FET.

ELIGIBILITY:
Inclusion Criteria:

* Endometrial thickness ≥ 7 mm on the day of starting progesterone-based luteal phase support (LPS)
* Serum progesterone levels <1.5 ng/ml on the day of starting progesterone-based LPS
* LPS with micronized progesterone 400mg b.i.d.
* Regular cycles (>24 days, ≤ 38 days)
* IVF/ICSI with donated oocytes
* Single blastocyst stage embryo transfer
* First or second embryo transfer from the same cohort

Exclusion Criteria:

* Use of exogenous ovarian stimulation during FET
* Untreated hydrosalpinx, polyp, submucous myomas or severe adenomyosis
* Recurrent pregnancy loss (≥ 3 previous pregnancy losses)
* Recurrent implantation failure with embryos from oocyte donation (≥ 3 previous failed embryo transfers)
* Personalized initiation of exogenous progesterone according to a previous endometrial receptivity assay test

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study group will include a prospectively recruited cohort of ovulatory patients undergoing their first or second FET attempt following oocyte donation in a natural proliferative phase protocol. The control group will include a retrospective cohort of ovulatory patients undergoing a natural cycle frozen embryo transfer following oocyte donation.
Sampling Method: Probability Sample
Enrollment: 530 (Estimated)
Dates: Start 2024-02-23 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of appointments needed before cycle scheduling | Up to three weeks
  Number of visits for cycle monitoring until embryo transfer scheduling

SECONDARY OUTCOMES:
Cycle duration until embryo transfer (days) | Up to four weeks
  Number of days since the first day of menstrual bleeding until the day of embryo transfer
Proportion of patients with low progesterone values on the day of embryo transfer | One day
  Percentage of patients with low serum progesterone levels on the day of embryo transfer
Human corionic gonadotropin (hCG) positive rate | 10-14 days after ET
  Proportion of patients with a positive hCG test
Miscarriage rate | Up to 20 weeks after ET
  Proportion of patients with spontaneous loss of an intra-uterine pregnancy prior to 22 completed weeks of gestational age
Ongoing pregnancy rate | 9-11 weeks after ET
  Proportion of patients with a pregnancy beyond the 11th week
Live birth rate | 40 weeks after ET
  Proportion of patients with a live birth

OTHER OUTCOMES:
Serum Relaxin-2 levels | 5 weeks
  Serum Relaxin-2 levels (colateral study)
Serum Luteinizing Hormone (LH) levels | 5 days
  Serum LH levels (colateral study)

CONTACTS AND LOCATIONS:
Overall Officials: Ana R Neves, MP, Principal Investigator — Instutito Valenciano de Infertilidade de Lisboa (IVI-RMA Lisboa)
Locations (1):
- Instituto Valenciano de Infertilidade, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: Undecided